CLINICAL TRIAL: NCT05700851
Title: Effect of Immuno-nutrition on Systemic Inflammation in People Receiving Haemodialysis: a Pilot Study
Brief Title: Immuno-nutrition Supplementation in Haemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21085; 309937 (Other: IRAS ID)
Record Dates: First submitted 2022-09-05; First posted 2023-01-26 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Haemodialysis; Systemic inflammation; Skeletal muscle mass; Immuno-nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immuno-nutrition (Other): Participants will be advised to take daily one sachet (74 g) of the immuno-nutrition supplement (Oral Impact®, Nestle) dissolved in 125 ml of water and will be followed-up for 6 weeks.
  Participants will receive individualised (to patient needs and food preferences) dietetic advice formulated and delivered by an experienced renal dietitian under an honorary NHS research contract, who is a member of the research team and will be supervised by an NHS renal dietitian, aiming to achieve estimated nutritional requirements for people on haemodialysis (i.e., energy: 30-35 kcal/kg/day, and protein intake: 1.0-1.2 g/kg/day). Each dietetic advice provided to participants will also be reviewed by the NHS clinical renal dietitians who are members of the participants' usual clinical care team.
  Interventions: Dietary Supplement: Immuno-nutrition supplement

INTERVENTIONS:
Dietary Supplement: Immuno-nutrition supplement — Oral Impact® is a powdered oral nutritional supplement that contains a unique combination of ingredients with immuno-modulating properties, namely omega-3 fatty acids, arginine and nucleotides, as well as soluble fibre.
  Other Names: Oral Impact®, Nestlé

SUMMARY:
The purpose of this pilot study is to test if an "immuno-nutrition" supplement can decrease inflammation in people on haemodialysis. This immuno-nutrition supplement is high in calories and protein like other common nutritional supplements, but also contains a unique combination of ingredients that have been shown to reduce inflammation (a problem which is caused by the body's defence [immune] system communicating that something is wrong) and improve the immune system in people with cancer. The research team hopes that this small study will help with gaining a good understanding of the effect of immuno-nutrition on inflammation in people on haemodialysis, which will guide and allow the research team to do a larger research study in the future.

DETAILED DESCRIPTION:
Participants will be asked to take one sachet of the immuno-nutrition supplement each day for 6 weeks. The renal dietitian on the research team will provide participants with detailed oral advice on how and when to take the immuno-nutrition supplement.

Participants will need to complete 3-day food diaries at the beginning, mid-way point and end of the study.

The research team will measure weight, height, handgrip strength (a measure of muscle strength), body's composition of fat and muscle using a specialist scale, and skin autofluorescence levels (a measure of toxins called advanced glycation end-products).

The research team will collect the results of routine blood tests. The research team will also collect and store blood samples taken before and after a haemodialysis session to measure some molecules that indicate inflammation.

All of these measurements and samples will be taken at the start of the study, and after 6 weeks of taking the immuno-nutrition supplement.

ELIGIBILITY:
Inclusion Criteria:

* CRP level >5.0 mg/L.
* At least three haemodialysis sessions per week for ≥3 hours using a biocompatible dialyser.
* Able to give informed consent.

Exclusion Criteria:

* Treatment with drugs that cause immunosuppression.
* Non-English speakers or those with special communication needs.
* Pregnancy, breast feeding or intending pregnancy.
* Expected survival <6 months.
* Hospitalisation at the time of screening.
* Known intolerance or allergy to ONS (or isolated ingredients).
* Pre-dialysis serum potassium >5.0 mmol/L.
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Taal, Principal Investigator — University of Nottingham
Locations (1):
- Department of Renal Medicine, Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Immuno-nutrition: Participants will be advised to take daily one sachet (74 g) of the immuno-nutrition supplement (Oral Impact®, Nestle) dissolved in 125 ml of water and will be followed-up for 6 weeks.
  Participants will receive individualised (to patient needs and food preferences) dietetic advice formulated and delivered by an experienced renal dietitian under an honorary NHS research contract, who is a member of the research team and will be supervised by an NHS renal dietitian, aiming to achieve estimated nutritional requirements for people on haemodialysis (i.e., energy: 30-35 kcal/kg/day, and protein intake: 1.0-1.2 g/kg/day). Each dietetic advice provided to participants will also be reviewed by the NHS clinical renal dietitians who are members of the participants' usual clinical care team.
  Immuno-nutrition supplement: Oral Impact® is a powdered oral nutritional supplement that contains a unique combination of ingredients with immuno-modulating properties, namely omega-3 fatty acids, arginine and nucleotides, as well as soluble fibre.
Period: Overall Study
Arm/Group | Immuno-nutrition
Started | 17
Completed | 14
Not Completed | 3
Not completed — Received a kidney transplant | 1
Not completed — Hospitalisation before starting baseline assessments | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Immuno-nutrition
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
C reactive protein [Median (Inter-Quartile Range); unit: mg/L] | 7.6 [4.8 to 32.3]
Interleukin-6 [Median (Inter-Quartile Range); unit: pg/mL] | 15.3 [7.0 to 22.4]
Interleukin-8 [Median (Inter-Quartile Range); unit: pg/mL] | 7.0 [2.4 to 9.5]
Handgrip strength [Median (Inter-Quartile Range); unit: kg] | 23.8 [17.1 to 27.9]
Skeletal muscle mass [Median (Inter-Quartile Range); unit: kg] | 26.7 [25.3 to 33.6]
Energy intake [Median (Inter-Quartile Range); unit: kcal/kg of body weight/day] | 26.6 [22.5 to 33.8]
Protein intake [Median (Inter-Quartile Range); unit: g/kg of body weight/day] | 1.0 [0.9 to 1.3]

OUTCOME MEASURES:

1. Primary Outcome: C Reactive Protein - Marker of Systemic Inflammation
Description: C reactive protein levels in mg/L using a high-sensitive laboratory test
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Immuno-nutrition
Number analyzed (Participants) | 14
mg/L | 7.3 [2.9 to 22.0]

2. Primary Outcome: Interleukin-6 - Marker of Systemic Inflammation
Description: Interleukin-6 levels in pg/ml using enzyme-linked immunosorbent assay
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Immuno-nutrition
Number analyzed (Participants) | 14
pg/mL | 10.5 [8.4 to 25.0]

3. Primary Outcome: Interleukin-8 - Marker of Systemic Inflammation
Description: Interleukin-8 levels in pg/ml using enzyme-linked immunosorbent assay
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Immuno-nutrition
Number analyzed (Participants) | 14
pg/mL | 4.9 [2.2 to 7.8]

4. Secondary Outcome: Skeletal Muscle Mass
Description: Skeletal muscle mass in kg assessed with the InBody 770 Multi-Frequency Bioimpedance Analysis equipment.
Time Frame: 6 weeks
Population: Skeletal muscle mass assessment requires participants to stand in the InBody equipment; therefore, skeletal muscle mass was not measured in 2 participants due to leg amputations. A contraindication for using the InBody equipment is having body metal implants; therefore, skeletal muscle mass was not measured in 1 participant due to this reason.
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Immuno-nutrition
Number analyzed (Participants) | 11
kg | 26.7 [23.9 to 32.3]

5. Secondary Outcome: Energy Intake
Description: Energy intake in kcal/kg of body weight/day assessed with 3-day food diaries and analysed using the diet software Nutritics
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: kcal/kg of body weight/day
Arm/Group | Immuno-nutrition
Number analyzed (Participants) | 14
kcal/kg of body weight/day | 27.2 [22.3 to 31.6]

6. Secondary Outcome: Protein Intake
Description: Protein intake in g/kg of body weight/day assessed with 3-day food diaries and analysed using the diet software Nutritics
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: g/kg of body weight/day
Arm/Group | Immuno-nutrition
Number analyzed (Participants) | 14
g/kg of body weight/day | 1.1 [1.0 to 1.4]

7. Secondary Outcome: Handgrip Strength - a Measure of Muscle Strength
Description: Handgrip strength in kg measured with the Takei 5401 handgrip digital dynamometer
Time Frame: 6 weeks
Population: Handgrip strength was not measured in 2 participants due to arthritis
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Immuno-nutrition
Number analyzed (Participants) | 12
kg | 24.4 [18.9 to 30.8]

ADVERSE EVENTS:
Time Frame: Reporting/recording of adverse event data was conducted from the baseline assessment until the end of the 6-week intervention period.
Arm/Group | Immuno-nutrition
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immuno-nutrition (N=16)
Intolerance to the immuno-nutrition supplement (Gastrointestinal disorders) | 1 (1) — Participant reported vomiting and diarrhoea after 4 days of taking the immuno-nutrition supplement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT05700851/Prot_SAP_000.pdf